CLINICAL TRIAL: NCT01960712
Title: The Role of Transpapillary Stenting in the Treatment of Bile Leakage After Liver Transection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Jansson, Anders, M.D. (Individual)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006/1142-31/3; 2006/1142-31/3 (Other: 2006/1142-31/3)
Record Dates: First submitted 2013-09-09; First posted 2013-10-11 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Bile Leakage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continued external drainage (No Intervention): Continued external drainage alone.
- Continued external drainage + transpapillary stent (Active Comparator): External drainage + transpapillary plastic stent (7-10 Fr).
  Interventions: Device: Transpapillary plastic stent (7-10 Fr)

INTERVENTIONS:
Device: Transpapillary plastic stent (7-10 Fr) — Duodenoscopy plus transpapillary bile cannulation plus stent insertion.
  Arms: Continued external drainage + transpapillary stent

SUMMARY:
Bile leakage after liver transection is treated by external drainage. The question addressed is whether downstream control by transpapillary stent insertion into distal bile duct can enhance healing.

DETAILED DESCRIPTION:
All patients who present with clinically significant bile leakage after liver resection at postoperative day two or longer are offered the opportunity to become randomized to either continuous external drainage or the addition of transpapillary stent.

ELIGIBILITY:
Inclusion Criteria:

* Liver resection including at least two liver segments.

Exclusion Criteria:

* Hepatobiliary digestive anastomosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of days of bile leakage from the abdominal cavity | From intervention until day discharge from hospital

SECONDARY OUTCOMES:
General complications rates. Postoperative hospital stay | From intervention until day of discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden